CLINICAL TRIAL: NCT04972643
Title: Department of Psychiatry, Taichung Veterans General Hospital
Brief Title: The Protective Effect of Omega-3 Fatty Acid on Cognitive Function Among Patients With Mild Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Tsuo-Hung Lan, Department of Psychiatry, Taichung Veterans General Hospital, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SF12109A
Record Dates: First submitted 2018-02-08; First posted 2021-07-22 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer Disease; Dementia Disorder
Keywords: Dementia Alzheimer
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EPA and DHA intervention (Experimental): EPA 1000mg and DHA 1000mg capsule twice a day, the total exposure to the intervention for each subject is 24 months.
  Interventions: Dietary Supplement: EPA; Dietary Supplement: DHA
- EPA intervention (Experimental): EPA 2000mg capsule twice a day, the total exposure to the intervention for each subject is 24 months.
  Interventions: Dietary Supplement: EPA
- DHA intervention (Experimental): DHA 2000mg capsule twice a day, the total exposure to the intervention for each subject is 24 months.
  Interventions: Dietary Supplement: DHA
- Placebo (Placebo Comparator): Placebo 2000mg capsule twice a day, the total exposure to the intervention for each subject is 24 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EPA — EPA 2000mg Soft capsules
  Arms: EPA and DHA intervention; EPA intervention
Dietary Supplement: DHA — DHA 2000mg Soft capsules
  Arms: DHA intervention; EPA and DHA intervention
Dietary Supplement: Placebo — Placebo Soft capsules
  Arms: Placebo

SUMMARY:
Background： Dementia is a progressive, devastating, and fatal neurodegenerative disorder. Alzheimer's disease (AD) is the most common cause of dementia, accounting for more than 50% of patients with dementia. Docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA), the major bioactive components of n-3 polyunsaturated fatty acids (n-3 PUFAs) , might connect to the etiology of several neuropsychiatric diseases. To our knowledge, it has never been studied to look at the different effects of DHA, EPA and their combination on associated symptoms of AD.

Objectives To examine the effects of DHA, EPA and their combination on associated symptoms of AD, including cognitive function, depressive symptoms, and functional ability.

Method This is a randomized, double-blind, placebo-controlled, 24-month follow-up study, enrolling 200-400 patients with mild AD (Mini-Mental Status Examination (MMSE) 19-26 or Clinical Dementia Rating (CDR) 0.5-1). Cognitive ability is assessed by the Alzheimer Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) and the MMSE. Mood status is assessed by Geriatric Depression Scale (GDS). Functional ability is assessed by the Alzheimer Disease Cooperative Study activities of daily living (ADCS-ADL) and global function by the CDR, quality of life scale (QOL-AD). Brain function is assessed by resting state brain magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Background Dementia is a progressive, devastating, and fatal neurodegenerative disorder (Cummings, 2004). As of 2010, there are an estimated 35.6 million people with dementia worldwide. By 2050, it is projected that this figure will have increased to over 115 million (1, 2). Therefore, dementia is not only an important medical disease but also a public health issue to demand immediate attention. A conservative estimate of economic burden from dementia (based on Alzheimer's Society's Dementia United Kindom (UK) report published in February 2007) reaches 20 billion by the year 2010, which suggests an average cost of 25,472 per person annually. It indicated a heavy social financial expense for the whole world in general. Alzheimer's disease (AD) is the most common cause of dementia, accounting for 60-80% of patients with dementia. Given that it is still lacking in effective treatments for AD, there has been growing interest in early detection and prevention for this disastrous illness. Delaying AD onset by 1 year could potentially lower its incidence by more than 9 million cases over the next 40 years (3).

Dementia could be resulted from numerous risk factors and medical conditions including vascular risk factors (e.g. hypertension, diabetes, and obesity), psychosocial factors (e.g. depression), and health behaviors (e.g. physical inactivity and smoking) (4, 5). Indeed, reflecting its heterogeneity, several hypotheses have been proposed for etiology of dementia, including genetic susceptibility, vascular changes, inflammatory process, oxidative stress, and recently, n-3 polyunsaturated fatty acids (n-3 PUFAs) (Fratiglioni et al., 2008;Samieri et al., 2008;Cole and Frautschy, 2010;Mucke and Pitas, 2004;Gomez-Pinilla, 2008). PUFAs are classified into mainly n-3 (or omega-3) and n-6 (or omega-6) groups. Docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA), the major bioactive components of n-3 PUFAs, are associated with neuronal membrane stability and fluidity, neurogenesis, neuroplasticity, neurotransmission and anti-inflammation, which might connect to the etiology of several neuropsychiatric diseases including depression and dementia (Horrobin and Bennett, 1999;Su et al., 2000;Chalon, 2006;Lukiw and Bazan, 2006;Su, 2009b;Lin et al., 2010a). On the other hand, arachidonic acid (AA), the major components of n-6 PUFAs, is a precursor of eicosanoids and is important to modulate proinflammatory effects, which might also link to the pathogenesis of neuroinflammatory and neurodegenerative diseases like dementia (Sanchez-Mejia and Mucke, 2010;Lukiw and Bazan, 2010). Consistent with the theoretical relevance, evidences to link PUFAs to dementia have been reported extensively from more epidemiological studies. For example, it has been observed that regions with a high consumption of fish, which are good sources of n-3 PUFAs, appear to have a lower prevalence of dementia (Barberger-Gateau et al., 2002;Barberger-Gateau et al., 2007;Huang et al., 2005;Morris et al., 2003;Kalmijn et al., 1997) and Mild cognitive Impairment (MCI) ;(Roberts et al., 2010)). Although clinical studies until now have failed to demonstrate beneficial effects of n-3 PUFA supplementation in patients with moderate or severe AD (Freund-Levi et al., 2006a;Quinn et al., 2010a), it may benefit in patients with mild AD or MCI and those without apolipoprotein E(APOE) ε4 allele (Freund-Levi et al., 2006b;Chiu et al., 2008;Quinn et al., 2010b). In addition, the two main n-3 PUFAs have different biological effects. DHA is the main n-3 PUFAs in the brain and is important in neuroplasticity and neuroprotection. EPA, on the other hand, is very little in the brain but is important in modulate inflammation and immune function (Lin et al., 2010b;Su, 2009a). To our knowledge, it has never been studied to look at the different effects of DHA, EPA and their combination on different associated symptoms of AD. To provide more evidence for the association between n-3 PUFAs and associated symptoms of AD, including cognitive function, depression, and physical activity in AD, we propose to conduct this double-blind, placebo-controlled, 24-month research. In addition, neuroprotective effects of vitamin B, preliminary findings in recent studies have shown cognitive-protection effects of it among patients with MCI. Moreover, deficiency of vitamin B is known to cause nervousness, depression, and peripheral and central neuropathy. The importance of vitamin B in developmental processes of the brain is supported by the findings that vitamin B deficiency at certain stages of brain development interferes with brain cell proliferation, migration and maturation . Vitamin B affords survival-promoting activities on cultured brain neurons (6). This is probably the first study to evaluate the effects of vitamin B on cognitive protection among Asian patients with AD. Based on the review of the possible benefits from n-3 PUFAs supplement on cognitive function preservation after balancing for its slightest side effects, we here propose a randomized clinical trial study design to test whether Hypothesis Omega-3 PUFAs is protective against cognitive decline among people with mild AD.

Primary Aim To examine whether consumption of n-3 PUFAs protects against cognitive decline in patients with mild AD.

Secondary Aims

1. To examine the different effects of DHA, EPA and their combination on different symptoms of AD.
2. To examine whether consumption of n-3 PUFAs improves cognitive function in patients with mild AD.
3. To examine whether consumption of n-3 PUFAs improves depressive symptoms in patients with mild AD.
4. To examine whether consumption of n-3 PUFAs improves physical activity level in patients with mild AD.

Significance of Study

1. To provide a simple way through dietary supplement of n-3 PUFAs to prevent cognitive decline and improve depressive symptoms and physical activity in patients with mild AD.
2. No placebo-controlled studies regarding n-3 PUFAs in cognitive prevention have been conducted among Asian people.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be included in the study if they meet the following criteria:

  1. Males and females over 65 years of age.
  2. Diagnosis of Alzheimer's Dementia disorder.
  3. Each individual must have a level of understanding sufficient to perform all tests and examinations required.
  4. Individuals must be willing to accept all laboratory examinations and MRI examination.
  5. Individuals must be willing to provide a small sample of blood for evaluation.
  6. Individuals must be willing to participate in a short 30-60 minute clinical interview.

Exclusion Criteria:

* Patients may be excluded from the study for any of the following reasons:

  1. Serious unstable illness such that death is anticipated within 1 year or intensive care unit hospitalization for the condition is anticipated within 6 months.
  2. Diagnosis of Vascular Dementia disorder.
  3. Uncorrected hypothyroidism or hyperthyroidism
  4. Participants will be excluded if they had evidence of epilepsy; focal brain lesion; head injury with loss of consciousness or confusion after the injury; DSMIV-TR (text revision) criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, or alcohol or substance abuse; or potential bleeding tendency.
  5. History of allergy to fish or omega-3 polyunsaturated fatty acids.

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-09-23 (Actual); Primary Completion 2018-05-12 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Aspartate Aminotransferase (AST) | Day 0
Aspartate Aminotransferase (AST) | Day 24 month
Alanine Aminotransferase (ALT) | Day 0
Alanine Aminotransferase (ALT) | Day 24 month
Albumin level | Day 0
Albumin level | Day 24 month
Fasting blood glucose | Day 0
Fasting blood glucose | Day 24 month
Blood Urea Nitrogen (BUN) | Day 0
Blood Urea Nitrogen (BUN) | Day 24 month
Creatinine level | Day 0
Creatinine level | Day 24 month
Sodium (Na) | Day 0
Sodium (Na) | Day 24 month
Potassium (K) | Day 0
Potassium (K) | Day 24 month
Calcium (Ca) | Day 0
Calcium (Ca) | Day 24 month
Magnesium (Mg) | Day 0
Magnesium (Mg) | Day 24 month
Triiodothyronine (T3) | Day 0
Triiodothyronine (T3) | Day 24 month
Free tetraiodothyronine (free T4) | Day 0
Free tetraiodothyronine (free T4) | Day 24 month
Thyroxin stimulating hormone (TSH) | Day 0
Thyroxin stimulating hormone (TSH) | Day 24 month
Triglycerides | Day 0
Triglycerides | Day 24 month
Total cholesterol | Day 0
Total cholesterol | Day 24 month
High density lipoprotein cholesterol (HDL) | Day 0
High density lipoprotein cholesterol (HDL) | Day 24 month
Low density lipoprotein cholesterol (LDL) | Day 0
Low density lipoprotein cholesterol (LDL) | Day 24 month
Vitamine B12 level | Day 0
Vitamine B12 level | Day 24 month
Folic acid | Day 0
Folic acid | Day 24 month
Rapid plasma reagin for Syphilis test (RPR) | Day 0
Rapid plasma reagin for Syphilis test (RPR) | Day 24 month
Mini Mental Status Evaluation (MMSE) total score | Day 0
  Minimu:0, Maximum: 30, Higher scores mean a better outcome.
Mini Mental Status Evaluation (MMSE) total score | Day 24 month
  Minimu:0, Maximum: 30, Higher scores mean a better outcome.
Clinical Dementia Rating Scale (CDR) total score | Day 0
  Minimu:0, Maximum: 3, Higher scores mean a worse outcome.
Clinical Dementia Rating Scale (CDR) total score | Day 24 month
  Minimu:0, Maximum: 3, Higher scores mean a worse outcome.
Hachinski ischemic score total score | Day 0
  Minimu:0, Maximum: 18, Higher scores mean a worse vascular outcome.
Hachinski ischemic score total score | Day 24 month
  Minimu:0, Maximum: 18, Higher scores mean a worse vascular outcome.
Alzheimer's Disease Assessment Scale-cognitive section (ADAS-Cog) total score | Day 0
  Minimu:0, Maximum: 70, Higher scores mean a worse outcome.
Alzheimer's Disease Assessment Scale-cognitive section (ADAS-Cog) total score | Day 24 month
  Minimu:0, Maximum: 70, Higher scores mean a worse outcome.
Alzheimer's Disease Assessment Scale-activities of daily living section (ADCS-ADL) total score | Day 0
  Minimu:0, Maximum: 54, Higher scores mean a better outcome.
Alzheimer's Disease Assessment Scale-activities of daily living section (ADCS-ADL) total score | Day 24 month
  Minimu:0, Maximum: 54, Higher scores mean a better outcome.
Geriatric Depression Scale (GDS) total score | Day 0
  Minimu:0, Maximum: 15, Higher scores mean a worse outcome.
Geriatric Depression Scale (GDS) total score | Day 24 month
  Minimu:0, Maximum: 15, Higher scores mean a worse outcome.
Quality of Life- Alzheimer Dementia (QOL-AD) total score | Day 0
  Minimu:13, Maximum: 52, Higher scores mean a better outcome.
Quality of Life- Alzheimer Dementia (QOL-AD) total score | Day 24 month
  Minimu:13, Maximum: 52, Higher scores mean a better outcome.
MRI examination 1 | Day 0
  Total brain volume: MRI examination will be performed on the 1.5 Telsla machine (GE, USA)
MRI examination 2 | Day 24 months
  Total brain volume: MRI examination will be performed on the 1.5 Telsla machine (GE, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Tsuo-Hung Lan, MD, PhD., Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- Taichung Veterans General Hospital, Taichung, No.450,Sec.1,Dongda Rd.,Xitun Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferri CP, Prince M, Brayne C, Brodaty H, Fratiglioni L, Ganguli M, Hall K, Hasegawa K, Hendrie H, Huang Y, Jorm A, Mathers C, Menezes PR, Rimmer E, Scazufca M; Alzheimer's Disease International. Global prevalence of dementia: a Delphi consensus study. Lancet. 2005 Dec 17;366(9503):2112-7. doi: 10.1016/S0140-6736(05)67889-0. PMID 16360788
- [Background] World Alzheimer Report 2010. Alzheimer's Disease International, 2010.
- [Background] Brookmeyer R, Johnson E, Ziegler-Graham K, Arrighi HM. Forecasting the global burden of Alzheimer's disease. Alzheimers Dement. 2007 Jul;3(3):186-91. doi: 10.1016/j.jalz.2007.04.381. PMID 19595937
- [Background] Daviglus ML, Bell CC, Berrettini W, Bowen PE, Connolly ES Jr, Cox NJ, Dunbar-Jacob JM, Granieri EC, Hunt G, McGarry K, Patel D, Potosky AL, Sanders-Bush E, Silberberg D, Trevisan M. National Institutes of Health State-of-the-Science Conference statement: preventing alzheimer disease and cognitive decline. Ann Intern Med. 2010 Aug 3;153(3):176-81. doi: 10.7326/0003-4819-153-3-201008030-00260. Epub 2010 Jun 14. PMID 20547888
- [Background] Barnes DE, Yaffe K. The projected effect of risk factor reduction on Alzheimer's disease prevalence. Lancet Neurol. 2011 Sep;10(9):819-28. doi: 10.1016/S1474-4422(11)70072-2. Epub 2011 Jul 19. PMID 21775213
- [Background] Wang XD, Kashii S, Zhao L, Tonchev AB, Katsuki H, Akaike A, Honda Y, Yamashita J, Yamashima T. Vitamin B6 protects primate retinal neurons from ischemic injury. Brain Res. 2002 Jun 14;940(1-2):36-43. doi: 10.1016/s0006-8993(02)02587-8. PMID 12020872